CLINICAL TRIAL: NCT04081974
Title: Prevalence and Predictors of Distal Limb Ischemia in Minimally Invasive Cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Other Study IDs: Leg perfusion
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Perfusion; Complications
Keywords: Minimally invasive cardiac surgery; Distal limb perfusion; Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minimally invasive cardiac surgery: All consecutive patients presenting for minimally invasive cardiac surgery will be screened for participation to the study.
  Interventions: Other: Distal leg perfusion

INTERVENTIONS:
Other: Distal leg perfusion — On arrival in the operating room, oximeter pads of a NIRO-200NX (NIRO,Hamamatsu® , Japan) NIRS monitor will be placed on the muscles of the calf bilaterally. Lower extremity NIRS is an added monitoring tool as it is currently not being used in our institutional clinical management. Neither anesthetic nor surgical plans will be altered by the study and are left to the discretion of the attending consultant. Also, perfusion goals may not be altered to the results of the leg NIRS. Therefore, the NIRS display will be covered in the operating room throughout the surgery.

SUMMARY:
Peripheral arterial cannulation is a necessity for installation of cardiopulmonary bypass in minimally invasive cardiac surgery (MICS). In the vast majority of cases, the femoral artery is the preferred arterial cannulation site. Distal limb hypoperfusion and ischemia can occur in the cannulated limb since antegrade perfusion is not routinely provided. Furthermore, the diameter of the cannula required to maintain adequate cardiopulmonary bypass (CPB) flow is often approaching that of the patient's femoral artery diameter, compromising distal blood flow. The possibility of distal limb ischemia is often raised as a criticism to peripheral cannulation for cardiopulmonary bypass and by extent to minimally invasive cardiac surgery. Ischemia of the lower limb is of high incidence in patients undergoing extracorporeal membrane oxygenation (ECMO) therapy, in which the same femoral cannulation technique is used. Therefore this complication has extensively been described in ECMO literature. However, no clinical trials have been performed in patients undergoing MICS, despite the same cannulation and perfusion route. ECMO patients often differ from MICS patients in morbidity as well as in duration of cannulation. Up to now, one could not observe any clinical sequelae of limb ischemia in MICS patients but a formal study of distal leg perfusion in MICS is recommended to screen its safety and to identify possible risk factors.

DETAILED DESCRIPTION:
Study design and setting Single-center prospective observational cohort study in patients undergoing minimally invasive cardiac surgery with peripheral arterial cannulation. This is the standard of care in the institution of the investigators.

Population All consecutive patients presenting for minimally invasive cardiac surgery will be screened for participation to the study. Eligible participants fulfill all inclusion criteria and no exclusion criteria (described below in more detail).

NIRS Near infrared spectroscopy (NIRS) is currently accepted as the golden standard monitoring tool for tissue oxygenation and for early detection of ischemia. The NIRS measures and displays a percent regional oxygenation saturation (rSO2). This value quantifies the percentage of regional hemoglobin oxygen saturation. It is measured by an electrode placed on the skin, and is therefore totally non-invasive. NIRS originally has been used to measure brain saturation, but its indications have been extended to any region of interest. Multiple studies validated NIRS as a useful monitor for detection of ischemia of the lower extremities in various settings (ECMO patients, patients with peripherally vascular disease). Patton-Rivera at al. showed rSO2 differentials > 15% had a 100% sensitivity and specificity for the detection of clinically markable hypoperfusion of the cannulated leg in ECMO patients.

Data collection Patient demographics and medical history will be collected together with the EuroScore II i.e the estimated risk of in-hospital death after cardiac surgery. NIRS values will be coded and anonymously recorded onto a Universal Serial Bus (USB) device and saved on a pc with limited access. rSO2 differentials between the cannulated and non-cannulated leg and Tissue Oxygenation Index (TOI) differentials from baseline in the cannulated leg will be noted (%). After completion and publication of the study all data will be deleted from the device.

Data for analyses of variables will be extracted from the anesthetic and perfusion charts. These charts are stored in the patients individual record.

Interventions On arrival in the operating room, oximeter pads of a NIRO-200NX (NIRO,Hamamatsu® , Japan) NIRS monitor will be placed on the muscles of the calf bilaterally. Lower extremity NIRS is an added monitoring tool as it is currently not being used in our institutional clinical management. Neither anesthetic nor surgical plans will be altered by the study and are left to the discretion of the attending consultant. Also, perfusion goals may not be altered to the results of the leg NIRS. Therefore, the NIRS display will be covered in the operating room throughout the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing minimally invasive cardiac surgery older than 18 years.

Exclusion Criteria:

1. History of leg amputation.
2. Calf muscle atrophy due to neuromuscular disorder or muscle diseases.
3. Stanford type A aortic dissection.
4. BMI > 40.
5. Allergy for NIRS electrode.
6. Revision surgery < 72h after primary surgery.
7. Postoperative need for intra-aortic balloon pump and/or ECMO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting for minimally invasive cardiac surgery will be screened for participation to the study. Eligible participants fulfill all inclusion criteria and no exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Drop of 15% in regional oxygen saturation (rSO2) lasting 4 minutes or longer between the cannulated and non-cannulated limb | Duration of the surgery
  A drop of 15% or more in StO2 for ≥ 4 minutes between the cannulated and non-cannulated leg during the cannulation period

SECONDARY OUTCOMES:
Difference in tissue oxygenation index (TOI) compared to baseline | Duration of the surgery
  A TOI shift below 50% from baseline in the cannulated leg
Identification of predictors of poor distal perfusion in the cannulated limb | from surgery until 6 months after surgery
  Seven variables will be analyzed for correlation with elevated StO2 differentials to identify risk factors for distal limb ischemia after peripheral cannulation for CPB: Patient age, Patient sex, Previous artery disease, Type of surgery (coronary artery bypass graft vs valve surgery),Arterial cannula size, Duration of cannulation, Body Surface Area
Peripheral vascular surgery | 6 months after surgery
  Prevalence of peripheral vascular surgery within six months after cardiac surgery (telephonic follow-up after 6 months and revision of patients medical record)
Relationship between distal limb ischemia and acute kidney injury | through study completion, an average of 6 months
  Investigate a possible relationship between distal limb ischemia and acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No